CLINICAL TRIAL: NCT02601183
Title: Cranial Temperature, as an Early Diagnosis Marker for Hemorrhagic and Ischemic Stroke
Brief Title: Cranial Temperature Early Diagnose Hemorrhagic and Ischemic Stroke
Acronym: CTedHI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Tan Liang, Southwest hospital, Third Military Medical University
Other Study IDs: ThirdMMU-tl
Record Dates: First submitted 2015-11-07; First posted 2015-11-10 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
Keywords: brain temperture，thrombolysis，early diagnosis
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ischemic stroke: The patients in the group are diagnosed as ischemic stroke by CT or MRA examination within 8h following stroke attack.
- Hemorrhagic stroke: The patients in the group are diagnosed as hemorrhagic stroke by CT or MRA examination within 8h following stroke attack.

SUMMARY:
The cerebrovascular diseases can be approximately divided as two types, namely ischemic and hemorrhagic stroke. Intravenous thrombolysis within 3-4.5 hours is highly recommended for acute ischemic stroke patients. But it's difficult to diagnose the ischemic stroke with the hemorrhagic stroke from the early symptoms and signs. It's with high risk of enlarging the hematoma if the patients with hemorrhagic stroke received the thrombolytic drugs. And time cost by CT or MRI examination is likely to responsible for missing the narrow time window and poor prognosis of stroke patients. Consequently, seeking for a noninvasive, rapid, portable and inexpensive diagnosis method which can sensitively distinguish the stroke type before CT or MRI examination would be very helpful in treating the ischemic stroke patients.

Because of the blockage in the cerebral supply artery, the heat from circulatory system will sharply decrease in infracted hemisphere among the ischemic stroke patients. The reduced brain temperature influenced the temperature on the ipsilateral forehead according to the data of our animal and preliminary clinical trial. In contrast, the temperature of the ipsilateral hemisphere showed a mild increase among the ischemic stroke patients in our preliminary experiment. The difference of the temperature tendency on the ipsilateral forehead has a great chance to be an early physical mark.

In our study, 30 ischemic stroke patients and 30 hemorrhagic stroke patients will be recruited. In the process of recruitment, the patients with acute stroke attack in no more than 4.5 hours will be collected the temperature at the five point without head coverage, including ipsilateral tempora, ipsilateral forehead, galbella, contralateral forehead, and contralateral tempora. Then the stroke would be recruited into the ischemic and hemorrhagic group according to the later CT or MRI results in the hospital. The accuracy and sensibility of early brain temperature in distinguishing stroke type would be tested in comparison with the diagnosis of imaging examination.

DETAILED DESCRIPTION:
Stroke is the leading cause of morbidity and disability among the aged population around the world, and its incidence is still rising recently. The cerebrovascular diseases can be approximately divided as two types, namely ischemic and hemorrhagic stroke. Their pathophysiological processes and therapeutical strategies are totally different. For hemorrhagic stroke, which takes up about 20% patients with cerebrovascular diseases, there is a lack of valid medical management in the very early stage except surgical hematoma removal. Whereas it's the key management for ischemic stroke to recanalize the occluded artery and restore blood flow before the irreversible brain damage. According the Guidelines for the Prevention of Stroke in Patients with Stroke and Transient Ischemic Attack, intravenous thrombolysis within 3-4.5 hours is highly recommended for acute ischemic stroke patients. The time window of thrombolysis after ischemic stroke is extremely narrow and greatly affected the patients' outcomes.

Despite the efficacious therapy exists, the rate of successful early thrombolysis is still awfully low, especially in the developing countries. Only 3-5% stroke patients can take advantage of the early thrombolysis. There are two major reasons response for such a low successful thrombolysis rate, including the civilian and some first-aid personnel hasn't mastered the timing of thrombolysis therapy for ischemic stroke. That would be improved by propaganda and education of the stroke knowledge. But what's more critical is the difficulty to diagnose the ischemic stroke with the hemorrhagic stroke from the early symptoms and signs. It's with high risk of enlarging the hematoma if the patients with hemorrhagic stroke received the thrombolytic drugs. For this reason, it's hard for the doctors to provide the correct treatment at the first time before imaging examination finished. And the time cost by CT or MRI examination is likely to responsible for missing the narrow time window and poor prognosis of stroke patients. Consequently, seeking for a noninvasive, rapid, portable and inexpensive diagnosis method which can sensitively distinguish the stroke type before CT or MRI examination would be very helpful in treating the ischemic stroke patients. The new method would enable the first-aid personnel to judge the stroke type in the ambulance and decide to apply intravenous thrombolysis or not.

Because of the blockage in the cerebral supply artery, especially the cerebral middle artery which can't be compensated, the blood flow in the corresponding hemisphere would drop sharply among the ischemic stroke patients. Along with decreasing heat from circulatory system, the infracted hemisphere's temperature should drop. The reduced brain temperature influenced the temperature on the ipsilateral forehead according to the data of our animal and preliminary clinical trial. In contrast, the temperature of the ipsilateral hemisphere showed a mild increase among the ischemic stroke patients in our preliminary experiment. That's possibly because the early mitochondrial dysfunction and inflammatory reaction induced by the hematoma. The difference of the temperature tendency on the ipsilateral forehead has a great chance to be an early physical mark. Temperature test could be rapid and noninvasive, making this mark a promising method to help the doctors to distinguish the stroke type in very early stage. Earlier diagnosis of ischemic stroke means earlier thrombolysis and much better prognosis.

In our study, 30 ischemic stroke patients and 30 hemorrhagic stroke patients will be recruited. In the process of recruitment, the patients with acute stroke attack in no more than 4.5 hours will be collected the temperature at the five point without head coverage, including ipsilateral tempora, ipsilateral forehead, galbella, contralateral forehead, and contralateral tempora. Then the stroke would be recruited into the ischemic and hemorrhagic group according to the later CT or MRI results in the hospital. The accuracy and sensibility of early brain temperature in distinguishing stroke type would be tested in comparison with the diagnosis of imaging examination. It should be emphasized that the diagnosis and following treatment should depend on the imaging examination and our brain temperature test is rapid and noninvasive. The therapy of the recruited stroke patients wouldn't be influenced by the trial and should be as usual as the standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients aged 18 to 80 years. 2.Supratentorial hypertensive intracerebral hemorrhage diagnosed by head CT or MRI.

  3.The intracerebral hematoma is more than 10ml. 4.Ischemic stroke diagnosed by head CT or MRI. 5.Unilateral middle cerebral artery occlusion or infarcted volume more than 1/2 of a hemicerebrum.

  6.The head temperature collection within 4.5 hours following stroke attack. 7.Glasgow Coma Scale between 5-10.

Exclusion Criteria:

* 1.the time after stroke attack exceed 4.5 hours. 2.The intracerebral hematoma is less than 10ml. 3.The infarcted volume less than 1/3 of a hemicerebrum. 4.With terminal cerebral hernia. 5.Pregnant women. 6.Serious impaired liver function, coagulation disorders, AIDS, combine other tumor or special condition.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with a symptom and sign of acute stroke admitted to a specialized stroke service within 4.5 hours.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Diagnose accordance rate | 24 hours
  This evaluation will be based on how accordant ischemic stroke diagnosis by cranial temperature compared with imaging examination.

SECONDARY OUTCOMES:
Diagnose accordance rate | 14 days
  This evaluation will be based on how accordant ischemic stroke diagnosis by cranial temperature compared with later clinical diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- the Southwest hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637